CLINICAL TRIAL: NCT04523376
Title: Closely Matched Unrelated Donor Peripheral Blood Stem Cell Transplantation with TCRαβ+ T Cell and B Cell Depletion for Patients with Sickle Cell Disease and Thalassemia Major
Brief Title: Pilot Study PBSCT with TCRab Depletion for Hemoglobinopathies
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Timothy Olson (Other)
Responsible Party: Sponsor-Investigator, Timothy Olson, Attending Physician, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-017141
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Sickle Cell Disease; Thalassemia Major
MeSH Terms: conditions — Anemia, Sickle Cell; beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Sickle Cell Disease (Experimental): Patients with Sickle Cell Disease (SCD) will be given previously established, disease-specific chemotherapy based conditioning regimens prior to hematopoietic stem cell transplantation using TCRalpha/beta and B cell depleted peripheral blood stem cells from closely matched unrelated donors.
  Interventions: Device: CliniMACS
- Beta Thalassemias Major (Experimental): Patients with Beta Thalassemias Major (BTM) will be given previously established, disease-specific chemotherapy based conditioning regimens prior to hematopoietic stem cell transplantation using TCRalpha/beta and B cell depleted peripheral blood stem cells from closely matched unrelated donors.
  Interventions: Device: CliniMACS

INTERVENTIONS:
Device: CliniMACS — Peripheral blood stem cells from closely matched unrelated donors will be processed using the CliniMACS device to remove TCRalpha/beta T cells and B cells, in accordance with the Investigator Brochure and Technical Manual following the laboratory standard operating procedures (SOPs) and using aseptic technique

SUMMARY:
This is a single arm pilot study of peripheral stem cell transplantation (PSCT) with ex vivo t-cell receptor alpha beta+(TCRαβ+) T cell and cluster of differentiation 19+ beta (CD19+ B) cell depletion of unrelated donor (URD) grafts using the CliniMACS device in patients with sickle cell disease (SCD) and beta thalassemia major (BTM).

DETAILED DESCRIPTION:
This is a single arm pilot study of peripheral stem cell transplantation (PSCT) with ex vivo TCRαβ+ T cell and CD19+ B cell depletion of URD grafts using the CliniMACS device in patients with SCD and BTM. Apart from CliniMACS-based cell processing, PSCT will be performed according to current standards of care in the Children's Hospital of Philadelphia (CHOP) Cell Therapy and Transplant Section, including the use of a standard chemotherapy conditioning regimen and standard follow-up laboratory assessments. The study will determine efficacy of this strategy in terms of engraftment, rates of acute and chronic Graft versus Host Disease (GvHD), and one-year overall and event-free survival.

ELIGIBILITY:
Inclusion criteria

Severe Sickle Cell Disease

* Genotype: Hemoglobin SS, Hemoglobin SC, Hemoglobin SD, SOArab, or Hemoglobin SBeta thalassemia
* Must have at least one of the following disease manifestations
* Clinically symptomatic neurologic event (stroke) or any neurologic deficit lasting greater than 24 hours at any time prior to enrollment
* History of two or more episodes of vaso-occlusive events (VOE) per year in the 2 years preceding enrolment. Patients must be refractory to hydroxyurea, defined as developing VOE despite receiving hydroxyurea for at least 6 months. Patients who are intolerant of hydroxyurea may also be enrolled.

Vaso-occlusive events include:

* Acute chest syndrome
* Pain episodes requiring intravenous pain management and/or hospitalization
* Priapism
* Splenic sequestration (defined as a 2 g/dL drop in hemoglobin in the setting of an acutely enlarging spleen. This will be determined as part of clinical care and prior to the research)
* Administration of regular red blood cell (RBC) transfusion therapy, defined as receiving ≥ 8 RBC transfusions in the year preceding enrollment to prevent sickle cell-related complications of any kind per treating hematologist's judgment.

Beta Thalassemia Major

* Genotype: Confirmed Beta Thalassemia genotype by molecular genetic testing (May include E/Beta0 and Beta0/Beta+ genotypes)
* Must meet clinical diagnosis of transfusion-dependent thalassemia, defined as need for ≥ 8 RBC transfusions per year in the two years preceding study enrollment.

Exclusion criteria

* Patients who do not meet disease, organ or infectious criteria.
* Previous Hematopoietic stem cell transplant (HSCT)
* Patients with no suitable unrelated donor available. Patients with suitable fully matched related donor are also not eligible.
* Pregnant females. All females of childbearing potential must have negative pregnancy test.
* Participation in a clinical trial in which the patient receives an investigational drug must be discontinued prior to the time of initiation of transplant therapy. Specifically transplant chemotherapy should not begin until at least 3 half-lives after last use of the investigational drug.
* Severe RBC alloimmunization, defined as inability to receive packed RBC transfusion therapy due to anti-RBC antibodies. Patients with high titer anti-donor human leukocyte antigen (HLA) antibodies detected on screening may be enrolled if they are willing to undergo HLA antibody desensitization therapy.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of graft failure | Up to 1year post-transplantation
  Number of patients with primary graft failure (defined as no evidence of neutrophil engraftment by day +30 after stem cell infusion) and secondary graft failure (defined as ANC <500 for at least 7-10 days after initial engraftment occurs in the absence of known infection or drug-mediated suppression, and confirmed by hypocellular bone marrow biopsy and/or total donor chimerism percentage from blood or bone marrow < 10 percent)
Time to neutrophil engraftment | Up to 60 days post-transplantation
  Number of days to neutrophil engraftment (first day of ANC >500/µl for the first of 3 consecutive days)
Incidence of acute graft vs. host disease (GVHD) | Up to 100 days post-transplantation
  Number of patients with acute GvHD (graded according to the current guidelines for reporting by the Center for International Bone Marrow Transplant Registry)
Incidence of chronic graft vs. host disease (GVHD) | Up to three years post-transplantation
  Number of patients with Grade II-IV acute GVHD, Severe Grade III-IV acute GVHD, and Chronic Extensive GVHD

SECONDARY OUTCOMES:
Number of deaths due to treatment | Up to 100 days post-transplantation
  Number of deaths due to treatment
Probability of event-free survival (EFS) | Up to 1 year post-transplantation
  Number of patients without complications or events
Probability of overall survival (OS) | 1 year post-transplantation
  Number of patients with the following survival outcome: one-year overall survival (OS)
Incidence of viral reactivation and symptomatic viral infection | Up to 1 year post-transplantation
  Number of patients experiencing viral reactivation requiring therapy and symptomatic viral infections, including CMV, adenovirus, and EBV

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Olson, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No